CLINICAL TRIAL: NCT00003656
Title: Phase II Trial of Atragen and Interferon Alfa-2b in Patients With Advanced Renal Cell Carcinoma
Brief Title: Tretinoin Plus Interferon Alfa in Treating Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9804003327; NYWCCC-0498-209; NCI-V98-1490
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Interferon-alpha

ARMS (1):
- All subjects (Experimental): Weekly ATRA-IV with recombinant interferon alfa
  Interventions: Biological: recombinant interferon alfa; Drug: tretinoin liposome

INTERVENTIONS:
Biological: recombinant interferon alfa
Drug: tretinoin liposome

SUMMARY:
RATIONALE: Tretinoin may help kidney cancer cells develop into normal cells. Interferon alfa may interfere with the growth of cancer cells.

PURPOSE: Phase II trial to study the effectiveness of liposomal tretinoin plus interferon alfa in treating patients who have metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response in patients with metastatic renal cell carcinoma treated with tretinoin liposome and interferon alfa-2b.
* Determine the toxicity of this regimen in these patients.
* Study retinoic acid receptor expression on tissue obtained from selected patients who have tumor biopsies.

OUTLINE: This is a dose-escalation study of tretinoin liposome with concurrent individual dose escalation of interferon alfa-2b. (Phase I closed to accrual as of 9/24/03.)

Patients receive tretinoin liposome IV over 30 minutes once weekly and interferon alfa-2b subcutaneously on five consecutive days (M-F) for 8 weeks. Courses repeat every 8 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of tretinoin liposome until the maximum tolerated dose (MTD) has been determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined additional patients are accrued and treated at that dose. (Phase I closed to accrual as of 9/24/03.)

During the first 3 weeks of the study, patients receive interferon alfa-2b at weekly dose escalations. After week 3, patients continue at the highest acceptable dose level of interferon alfa-2b for the remainder of the study. (Phase I closed to accrual as of 9/24/03.)

Patients are followed at 30 days after the last treatment.

PROJECTED ACCRUAL: A total of 3-18 patients will be accrued into the phase I portion of this study (Phase I closed to accrual as of 9/24/03). A total of 14-25 patients will be accrued into the phase II portion of this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic renal cell carcinoma
* Bidimensionally measurable disease
* No active brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* More than 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3
* No coagulation disorders

Hepatic:

* Bilirubin less than 1.5 mg/dL
* SGOT and SGPT less than 112.5 IU/L each or less than 2.5 times upper limit of normal
* No clinically significant hepatic disease, including autoimmune hepatitis

Renal:

* Creatinine less than 2 mg/dL OR
* Creatinine clearance greater than 50 mL/min
* No clinically significant renal disease

Cardiovascular:

* No clinically significant cardiac disease
* No thrombophlebitis

Pulmonary:

* No severe debilitating pulmonary disease
* No pulmonary embolism

Other:

* No history of diabetes mellitus prone to ketoacidosis
* No known hypersensitivity to retinoids or retinoic acid derivatives or to interferon or any component of the injection for this study
* No thyroid abnormalities that hinder maintaining thyroid function at the normal range
* No severe infection
* No severe malnutrition
* No clinically significant retinal abnormalities
* No pre-existing psychiatric condition, especially depression or a history of severe psychiatric disorder
* No other concurrent malignancy except nonmelanoma skin cancer or curatively treated carcinoma in situ of the cervix
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 effective methods of contraception during and for 1 month after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No more than 1 prior biological response modifier therapy or immunotherapy

Chemotherapy:

* No more than 1 prior chemotherapy regimen

Endocrine therapy:

* No concurrent steroids

Radiotherapy:

* At least 4 weeks since prior radiotherapy

Surgery:

* At least 4 weeks since prior major surgery

Other:

* No prior retinoid therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 1999-01 (Actual); Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M. Nanus, MD, Study Chair — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York

REFERENCES:
- [Background] Goldberg JS, Vargas M, Rosmarin AS, Milowsky MI, Papanicoloau N, Gudas LJ, Shelton G, Feit K, Petrylak D, Nanus DM. Phase I trial of interferon alpha2b and liposome-encapsulated all-trans retinoic acid in the treatment of patients with advanced renal cell carcinoma. Cancer. 2002 Sep 15;95(6):1220-7. doi: 10.1002/cncr.10809. PMID 12216088
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://www.ncbi.nlm.nih.gov/pubmed/?term=12216088

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from between April 2002 and March 2005. Data are only available as a combined Arm/Group based on information contained in the study publication. No additional study data is available despite exhausting all efforts to locate the data.
Groups:
- Phase 1 Group: Weekly ATRA-IV (with three dose levels: 60, 75, and 90 mg/m2) with recombinant interferon alfa recombinant interferon alfa tretinoin liposome
- Phase 2 Group: Weekly ATRA-IV (dosage of 90 mg/m2) with recombinant interferon alfa recombinant interferon alfa tretinoin liposome
Period: Overall Study
Arm/Group | Phase 1 Group | Phase 2 Group
Started | 12 | 14
Completed | 12 | 13
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Data are only available as a combined Arm/Group based on information contained in the study publication. No additional study data is available despite exhausting all efforts to locate the data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 Group | Phase 2 Group | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Customized [Mean (Inter-Quartile Range); unit: years]
  Median age | 66.5 [42 to 79] | 61.1 [47 to 75] | 63.6 [42 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 7 | 10 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Prior nephrectomy [Count of Participants; unit: Participants]
  Yes prior nephrectomy | 12 | 12 | 24
  No prior nephrectomy | 0 | 2 | 2
Histology [Count of Participants; unit: Participants]
  Clear cell | 7 | 9 | 16
  Clear cell with sarcomatoid features | 1 | 4 | 5
  Papillary | 1 | 0 | 1
  Xp11 | 0 | 1 | 1
  Unclassified | 3 | 0 | 3
Number of patients with metastases at the time of diagnosis [Count of Participants; unit: Participants] | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Best Response as Measured by CT, Bone Scans, and Clinical Progression
Time Frame: After 8 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Group | Phase 2 Group
Number analyzed (Participants) | 12 | 14
Participants
  Complete Response | 1 | 0
  Minor Reponse | 0 | 1
  Partial Response | 1 | 3
  Stable Disease | 5 | 4
  Disease Progression | 5 | 6

2. Primary Outcome: Number of Subjects With Toxicity by Clinical Evaluation From First Dose to 30 Days After Last Dose
Time Frame: In 30 days after the last dose, an average of 1 year.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Group | Phase 2 Group
Number analyzed (Participants) | 12 | 14
Participants
  Fatigue : Grade 1 | 7 | 8
  Fatigue : Grade 2 | 5 | 4
  Fatigue : Grade 3 | 0 | 0
  Fatigue : Grade 4 | 0 | 0
  Skin : Grade 1 | 1 | 3
  Skin : Grade 2 | 0 | 0
  Skin : Grade 3 | 0 | 0
  Skin : Grade 4 | 0 | 0
  Xeroderma : Grade 1 | 11 | 5
  Xeroderma : Grade 2 | 0 | 0
  Xeroderma : Grade 3 | 0 | 0
  Xeroderma : Grade 4 | 0 | 0
  Constipation : Grade 1 | 5 | 4
  Constipation : Grade 2 | 0 | 0
  Constipation : Grade 3 | 0 | 0
  Constipation : Grade 4 | 0 | 0
  Cough : Grade 1 | 4 | 0
  Cough : Grade 2 | 2 | 0
  Cough : Grade 3 | 0 | 0
  Cough : Grade 4 | 0 | 0
  Anemia : Grade 1 | 3 | 2
  Anemia : Grade 2 | 1 | 5
  Anemia : Grade 3 | 2 | 0
  Anemia : Grade 4 | 0 | 0
  Anorexia : Grade 1 | 9 | 6
  Anorexia : Grade 2 | 2 | 2
  Anorexia : Grade 3 | 0 | 0
  Anorexia : Grade 4 | 0 | 0
  Neurologic : Grade 1 | 8 | 9
  Neurologic : Grade 2 | 3 | 1
  Neurologic : Grade 3 | 1 | 0
  Neurologic : Grade 4 | 0 | 0
  Diarrhea : Grade 1 | 5 | 4
  Diarrhea : Grade 2 | 0 | 0
  Diarrhea : Grade 3 | 0 | 0
  Diarrhea : Grade 4 | 0 | 0
  Nausea/vomiting : Grade 1 | 2 | 6
  Nausea/vomiting : Grade 2 | 2 | 1
  Nausea/vomiting : Grade 3 | 0 | 0
  Nausea/vomiting : Grade 4 | 0 | 0
  Altered mood : Grade 1 | 8 | 4
  Altered mood : Grade 2 | 0 | 0
  Altered mood : Grade 3 | 0 | 0
  Altered mood : Grade 4 | 0 | 0
  Leukopenia : Grade 1 | 2 | 2
  Leukopenia : Grade 2 | 2 | 1
  Leukopenia : Grade 3 | 3 | 0
  Leukopenia : Grade 4 | 0 | 0
  Fever : Grade 1 | 4 | 5
  Fever : Grade 2 | 1 | 0
  Fever : Grade 3 | 0 | 0
  Fever : Grade 4 | 0 | 0
  Renal : Grade 1 | 1 | 3
  Renal : Grade 2 | 1 | 0
  Renal : Grade 3 | 0 | 0
  Renal : Grade 4 | 0 | 0
  Liver : Grade 1 | 1 | 2
  Liver : Grade 2 | 0 | 0
  Liver : Grade 3 | 0 | 0
  Liver : Grade 4 | 0 | 0
  Thrombocytopenia : Grade 1 | 2 | 3
  Thrombocytopenia : Grade 2 | 0 | 0
  Thrombocytopenia : Grade 3 | 0 | 0
  Thrombocytopenia : Grade 4 | 0 | 0
  Infusion reaction : Grade 1 | 0 | 0
  Infusion reaction : Grade 2 | 0 | 1
  Infusion reaction : Grade 3 | 0 | 0
  Infusion reaction : Grade 4 | 0 | 0
  Pulmonary : Grade 1 | 0 | 1
  Pulmonary : Grade 2 | 0 | 0
  Pulmonary : Grade 3 | 0 | 1
  Pulmonary : Grade 4 | 0 | 0
  Nasal congestion : Grade 1 | 0 | 1
  Nasal congestion : Grade 2 | 0 | 0
  Nasal congestion : Grade 3 | 0 | 0
  Nasal congestion : Grade 4 | 0 | 0
  Hypotension : Grade 1 | 0 | 0
  Hypotension : Grade 2 | 0 | 1
  Hypotension : Grade 3 | 0 | 0
  Hypotension : Grade 4 | 0 | 0
  Cholesterol/TG : Grade 1 | 0 | 1
  Cholesterol/TG : Grade 2 | 0 | 0
  Cholesterol/TG : Grade 3 | 0 | 0
  Cholesterol/TG : Grade 4 | 0 | 0
  Bone pain : Grade 1 | 0 | 1
  Bone pain : Grade 2 | 0 | 0
  Bone pain : Grade 3 | 0 | 0
  Bone pain : Grade 4 | 0 | 0
  Other pain : Grade 1 | 0 | 5
  Other pain : Grade 2 | 0 | 0
  Other pain : Grade 3 | 0 | 0
  Other pain : Grade 4 | 0 | 0

3. Secondary Outcome: Change in Retinoic Acid Receptor Expression on Tissue as Measured by Number of Subjects With the Presence of Peripheral Blood Lymphocytes During the First and Fifth Dose
Time Frame: At baseline and 5th week
Population: Phase 1 portion at the RP2D of 90 mg/m2. 6 patients (12 in phase 1 w 6 at 75 mg/m2 and 6 at 90 mg/m2). This was not completed on the other 14 in phase 2 portion.
Measure: Count of Participants; unit: Participants
Groups:
- All Subjects: Weekly ATRA-IV with recombinant interferon alfa
  recombinant interferon alfa
  tretinoin liposome
Arm/Group | All Subjects
Number analyzed (Participants) | 6
Participants | 0

4. Secondary Outcome: Duration of Response (Progression-free Survival) as Measured by CT, Bone Scans, and Clinical Progression From Initiation of Therapy Until an Increase of ≥ 25% From the Smallest Sum of All Tumor Measurements Obtained During the Best Response
Time Frame: At 6 months and 12 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Group | Phase 2 Group
Number analyzed (Participants) | 12 | 14
Participants
  6 month | 5 | 7
  12 month | 4 | 3

ADVERSE EVENTS:
Description: Data are only available as a combined Arm/Group based on information contained in the study publication. No additional study data is available despite exhausting all efforts to locate the data.
Arm/Group | Phase 1 Group | Phase 2 Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/14
Other Adverse Events (participants affected / at risk) | 12/12 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Group (N=12) | Phase 2 Group (N=14)
Leukopenia (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 Group (N=12) | Phase 2 Group (N=14)
Fatigue - Grade 1 (General disorders) | 7 | 8
Fatigue - Grade 2 (General disorders) | 5 | 4
Constipation - Grade 1 (Gastrointestinal disorders) | 5 | 4
Cough - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Cough - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Anemia - Grade 1 (Blood and lymphatic system disorders) | 3 | 2
Anemia - Grade 2 (Blood and lymphatic system disorders) | 1 | 5
Anemia - Grade 3 (Blood and lymphatic system disorders) | 2 | 0
Anorexia - Grade 1 (Metabolism and nutrition disorders) | 9 | 6
Anorexia - Grade 2 (Metabolism and nutrition disorders) | 2 | 2
Skin - Grade 1 (Skin and subcutaneous tissue disorders) | 1 | 3
Xeroderma - Grade 1 (Skin and subcutaneous tissue disorders) | 11 | 5
Neurologic - Grade 1 (Nervous system disorders) | 8 | 9
Neurologic - Grade 3 (Nervous system disorders) | 1 | 0
Diarrhea - Grade 1 (Gastrointestinal disorders) | 5 | 4
Nausea/Vomiting - Grade 1 (Gastrointestinal disorders) | 2 | 6
Nausea/Vomiting - Grade 2 (Gastrointestinal disorders) | 2 | 1
Altered Mood - Grade 1 (Psychiatric disorders) | 8 | 4
Leukopenia - Grade 1 (Blood and lymphatic system disorders) | 2 | 2
Leukopenia - Grade 2 (Blood and lymphatic system disorders) | 2 | 1
Leukopenia - Grade 3 (Blood and lymphatic system disorders) | 2 | 0
Fever - Grade 1 (Immune system disorders) | 4 | 5 — Side effect of interferon
Fever - Grade 2 (Immune system disorders) | 1 | 0 — Side effect of interferon
Renal - Grade 1 (Renal and urinary disorders) | 1 | 3
Renal - Grade 2 (Renal and urinary disorders) | 1 | 0
Liver - Grade 1 (Hepatobiliary disorders) | 1 | 2
Thrombocytopenia - Grade 1 (Blood and lymphatic system disorders) | 2 | 3
Infusion Reaction - Grade 2 (General disorders) | 0 | 1
Pulmonary - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension - Grade 2 (Cardiac disorders) | 0 | 1
Cholesterol/TG - Grade 1 (Blood and lymphatic system disorders) | 0 | 1
Bone Pain - Grade 1 (Musculoskeletal and connective tissue disorders) | 0 | 1
Other Pain - Grade 1 (General disorders) | 0 | 5
Neurologic - Grade 2 (Nervous system disorders) | 3 | 1
Pulmonary - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal Congestion - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No